CLINICAL TRIAL: NCT04547023
Title: Fasting Versus Fed: Effect of Oral Intake Prior to the Glucose Tolerance Test in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Yair Blumenfeld, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 57772; P30DK116074 (NIH)
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Results first posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-10

CONDITIONS: Gestational Diabetes; Diagnoses Disease; Pregnancy in Diabetic; Glucose, High Blood
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy in Diabetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting before gestational diabetes screen (Experimental): Fasting for at least 6 hours prior to the 1-hour gestational diabetes screen.
  Interventions: Behavioral: Fasting before gestational diabetes screen
- Fed before gestational diabetes screen (Active Comparator): Liberal per oral intake within 2 hours of the 1-hour gestational diabetes screen.
  Interventions: Behavioral: Per oral intake of food and drink

INTERVENTIONS:
Behavioral: Fasting before gestational diabetes screen — Fasting for at least 6 hours before 1-hour gestational diabetes screen.
  Arms: Fasting before gestational diabetes screen
Behavioral: Per oral intake of food and drink — Per oral intake of food and drink within 2 hours of gestational diabetes screen
  Arms: Fed before gestational diabetes screen

SUMMARY:
Studies suggest that the timing interval between oral intake and the 1-hour gestational diabetes screen may have a significant impact on gestational diabetes screening glucose levels. The investigators plan to conduct a prospective randomized trial comparing a 6-hour fast versus liberal oral intake within 2 hours prior to the glucose tolerance test in pregnancy in order to evaluate the effect of the fasting versus the fed state on routine gestational diabetes screening results.

DETAILED DESCRIPTION:
Gestational diabetes (GDM) complicates approximately 400,000 pregnancies in the United States annually and is associated with significant adverse pregnancy outcomes, including increasing the lifetime risk of type 2 diabetes. The American College of Obstetricians and Gynecologists (ACOG) recommends that all pregnant women undergo GDM screening between 24-28 weeks gestation utilizing a 1-hour oral glucose tolerance test that was designed to be administered without regard to the last meal or time of day. However, studies suggest that the timing of one's last meal prior to the 1-hour GDM screen may have a significant impact on GDM screening glucose levels. In addition, providers routinely alter the timing of the 1-hour GDM screen based on patients' self reported oral intake prior to the exam. The investigators plan to conduct a prospective randomized trial comparing a 6-hour fast versus liberal oral intake within 2 hours prior to the glucose tolerance test in pregnancy in order to evaluate the effect of the fasting versus the fed state on routine GDM screening results.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant patients 18 years and older
2. Singleton gestation
3. Pregnancy managed at Lucile Packard Children's Hospital (LPCH) Stanford outpatient obstetrics clinic
4. Planned delivery at Lucile Packard Children's Hospital (LPCH) Stanford Labor and Delivery unit

Exclusion Criteria:

1. Pregestational diabetes
2. Gestational diabetes diagnosed in the 1st trimester
3. Less than 18 years of age
4. Planned delivery outside LPCH
5. Diabetes medication use prior to pregnancy
6. Inability to give informed consent
7. Chronic steroid use in pregnancy
8. Less than 24 weeks of gestation at the time of the 1 hour oral glucose tolerance test
9. Prior history of bariatric surgery
10. Multifetal gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yair Blumenfeld, MD, Principal Investigator — Associate Professor
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sperling MM, Leonard SA, Miller SE, Hurtado J, El-Sayed YY, Herrero T, Faig J, Carter S, Blumenfeld YJ. Fasting Compared With Fed and Oral Intake Before the 1-Hour Oral Glucose Tolerance Test: A Randomized Controlled Trial. Obstet Gynecol. 2023 Jan 1;141(1):126-133. doi: 10.1097/AOG.0000000000005013. Epub 2022 Nov 30. PMID 36701613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled pregnant participants. While outcomes were assessed in neonates, they were not considered to be enrolled.
Period: Overall Study
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Started | 100 | 100
Completed | 96 | 97
Not Completed | 4 | 3
Not completed — Did Not Receive Intervention | 3 | 2
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (4.2) | 33.2 (4.7) | 32.7 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 200
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/ Pacific Islander | 39 | 35 | 74
  Hispanic | 6 | 17 | 23
  Non-Hispanic Black | 2 | 3 | 5
  Non-Hispanic White | 49 | 40 | 89
  Other | 4 | 5 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Positive Gestational Diabetes Mellitus (GDM) Screen (>= 140 mg/dL) on the 1 Hour 50-g Oral Glucose Tolerance Test (OGTT)
Description: Number of positive GDM screen (>= 140 mg/dL) on the 1 hour 50-g oral glucose tolerance test conducted between 24-28 weeks gestation This outcome was assessed in pregnant participants.
Time Frame: Day of GDM screen (occurring between 24-28 weeks gestation)
Population: Participants who completed the 1 hour GDM screen are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 97 | 98
Participants | 31 | 13
Statistical Analysis 1: Comparison: Fasting Before Gestational Diabetes Screen vs Fed Before Gestational Diabetes Screen; Test type: Other; p = 0.002, Fisher Exact; Mean Difference (Final Values) = 18.7, 95% CI 2-sided [7.2 to 30.1]

2. Secondary Outcome: Mean Gestational Age at OGTT Screen
Time Frame: Day of GDM screen (occurring between 24-28 weeks gestation)
Population: Participants who completed the 1 hour GDM screen are included in the analysis
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 97 | 98
weeks | 25.7 (1.2) | 25.8 (1.3)

3. Secondary Outcome: Mean Glucose Level at the OGTT Screen
Time Frame: Day of GDM screen (occurring between 24-28 weeks gestation)
Population: Participants who completed the 1 hour GDM screen are included in the analysis
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 97 | 98
mg/dL | 127.7 (35.8) | 113.3 (26.4)

4. Secondary Outcome: Number of Participants With Positive GDM Diagnosis Based on the OGTT
Description: This outcome was assessed in pregnant participants.
Time Frame: Day of GDM screen (occurring between 24-28 weeks gestation)
Population: Participants who completed the 1 hour GDM screen are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 97 | 98
Participants | 8 | 2

5. Secondary Outcome: Average Time of Last Oral Intake Prior to the OGTT Screen
Description: Average number of hours since the participant's last oral intake prior to OGTT screen
Time Frame: Day of GDM screen (occurring between 24-28 weeks gestation)
Population: Participants who completed the 1 hour GDM screen are included in the analysis
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 97 | 98
hours | 10.7 (3.0) | 1.4 (0.9)

6. Secondary Outcome: Number of Participants With Positive GDM Diagnosis
Description: GDM diagnosis based on 1-hour OGTT ≥ 180 mg/dL or 2 elevated values on the 3-hour OGTT using Carpenter and Coustan criteria. This outcome was assessed in pregnant participants
  Carpenter and Coustan Criteria is as follows (if 2 or more values are elevated, this is gestational diabetes):
  * Fasting glucose < 95;
  * One hour glucose < 180;
  * Two hour glucose < 155;
  * Three hour glucose < 140
Time Frame: Day of OGTT (occurring at 24-28 weeks gestation up to 42 weeks gestation)
Population: Participants who completed the 1 hour GDM screen are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 97 | 98
Participants | 12 | 5

7. Secondary Outcome: Mean Gestational Age at Delivery
Time Frame: At time of delivery (Up to 42 weeks' gestation)
Population: Participants who had delivery data are included in the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 96
days | 272 (12) | 272 (10)

8. Secondary Outcome: Number of Participants Who Delivered Vaginally
Description: This outcome was assessed in pregnant participants.
Time Frame: At time of delivery (up to 42 weeks' gestation)
Population: Participants who had delivery data are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 96
Participants | 67 | 53

9. Secondary Outcome: Number of Participants Who Delivered Via Operative Vaginal Birth
Description: This outcome was assessed in pregnant participants.
Time Frame: At time of delivery (up to 42 weeks' gestation)
Population: Participants who had delivery data are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 96
Participants | 3 | 7

10. Secondary Outcome: Number of Participants Who Delivered Vaginally After a Prior Cesarean Section
Description: This outcome was assessed in pregnant participants.
Time Frame: At time of delivery (up to 42 weeks' gestation)
Population: Participants who had delivery data are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 96
Participants | 2 | 1

11. Secondary Outcome: Number of Participants Who Delivered Via a Primary Cesarean Section
Description: Primary = first Cesarean section for participant. This outcome was assessed in pregnant participants.
Time Frame: At time of delivery (up to 42 weeks' gestation)
Population: Participants who had delivery data are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 96
Participants | 17 | 21

12. Secondary Outcome: Number of Participants Who Delivered Via a Repeat Cesarean Section
Description: This outcome was assessed in pregnant participants.
Time Frame: At time of delivery (up to 42 weeks' gestation)
Population: Participants who had delivery data are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 96
Participants | 7 | 14

13. Secondary Outcome: Number of Participants Complicated by Shoulder Dystocia at Delivery
Description: Shoulder dystocia is a birth injury (also called birth trauma) that happens when one or both of a baby's shoulders get stuck inside the mother's pelvis during labor and birth. This outcome was assessed in pregnant participants.
Time Frame: At time of delivery (up to 42 weeks' gestation)
Population: Participants who had delivery data are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 96
Participants | 0 | 1

14. Secondary Outcome: Number of Participants Complicated by Third or Fourth Degree Perineal Laceration
Description: A third degree tear is a tear or laceration through the perineal muscles and the anal sphincter. A fourth degree tear goes through the anal sphincter all the way to the anal canal or rectum. This outcome was assessed in pregnant participants.
Time Frame: At time of delivery (up to 42 weeks' gestation)
Population: Participants who had delivery data are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 96
Participants | 2 | 4

15. Secondary Outcome: Number of Participants With Post-partum Hemorrhage
Description: This outcome was assessed in pregnant participants after delivery.
Time Frame: Up to 6 weeks after delivery
Population: Participants who had delivery data are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 96
Participants | 16 | 10

16. Secondary Outcome: Number of Participants Diagnosed With a Hypertensive Disorder of Pregnancy
Description: This outcome was assessed in pregnant participants.
Time Frame: From time of GDM screen up to 6 weeks after delivery
Population: Participants who had delivery data are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 96
Participants | 22 | 15

17. Secondary Outcome: Length of Postnatal Stay From Delivery to Discharge
Description: Average number of days admitted in the hospital after delivery up to discharge
Time Frame: Up to 1 week after delivery
Population: Participants who had delivery data are included in the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 96
days | 2.3 (0.9) | 2.4 (1.1)

18. Secondary Outcome: Number of Participants Who Had a Postpartum Readmission
Description: This outcome was assessed in pregnant participants post-delivery.
Time Frame: From initial hospital discharge up to 6 weeks post-partum
Population: Participants who had delivery data are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 96
Participants | 4 | 6

19. Secondary Outcome: Number of Participants With Type 2 Diabetes Mellitus Diagnosis Post-partum
Description: This outcome was assessed in pregnant participants after delivery.
Time Frame: From time of delivery up to 6 weeks post-partum
Population: Participants who had delivery data are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 96
Participants | 1 | 0

20. Secondary Outcome: Mean Neonatal Birthweight
Time Frame: Day of delivery (Within approximately 2 hours after delivery)
Population: Participants with a live birth are included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 95
grams | 3231 (631) | 3268 (458)

21. Secondary Outcome: Number of Neonates With Birth Weight More Than 4000 Grams
Time Frame: Day of delivery (Within approximately 2 hours after delivery)
Population: Participants with a live birth are included in the analysis.
Measure: Number; unit: neonates
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 95
neonates | 6 | 6

22. Secondary Outcome: Number of Neonates Considered Large for Gestational Age (LGA)
Description: LGA refers to neonatal birth weight larger than the 90th percentile for gestational age.
Time Frame: Day of delivery (Within approximately 2 hours after delivery)
Population: Participants with a live birth are included in the analysis.
Measure: Number; unit: neonates
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 95
neonates | 6 | 7

23. Secondary Outcome: Number of Neonates Considered Small for Gestational Age (SGA)
Description: SGA are infants whose weight is < the 10th percentile for gestational age.
Time Frame: Day of delivery (Within approximately 2 hours after delivery)
Population: Participants with a live birth are included in the analysis.
Measure: Number; unit: neonates
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 95
neonates | 6 | 9

24. Secondary Outcome: Number of Neonates Admitted to the Neonatal Intensive Care Unit (NICU)
Time Frame: Up to 28 days after delivery
Population: Participants with a live birth are included in the analysis.
Measure: Number; unit: neonates
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 95
neonates | 4 | 7

25. Secondary Outcome: Number of Neonates With Hyperbilirubinemia
Time Frame: Up to 28 days after delivery
Population: Participants with a live birth are included in the analysis.
Measure: Number; unit: neonates
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 95
neonates | 7 | 9

26. Secondary Outcome: Number of Neonates With Hypoglycemia
Time Frame: Up to 28 days after delivery
Population: Participants with a live birth are included in the analysis.
Measure: Number; unit: neonates
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 95
neonates | 9 | 5

27. Secondary Outcome: Number of Neonates Diagnosed With Respiratory Distress Syndrome
Time Frame: Up to 28 days after delivery
Population: Participants with a live birth are included in the analysis.
Measure: Number; unit: neonates
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 96 | 95
neonates | 7 | 7

28. Secondary Outcome: Number of Neonates Exclusively Breastfeeding at Time of Hospital Discharge
Time Frame: Up to 28 days after delivery
Population: Participants with breast feeding data are included in the analysis
Measure: Number; unit: neonates
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
Number analyzed (Participants) | 86 | 88
neonates | 62 | 59

ADVERSE EVENTS:
Time Frame: Up to 22 weeks (from 24 weeks gestation up to 6 weeks post-partum)
Arm/Group | Fasting Before Gestational Diabetes Screen | Fed Before Gestational Diabetes Screen
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 2/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fasting Before Gestational Diabetes Screen (N=100) | Fed Before Gestational Diabetes Screen (N=100)
Intrauterine fetal demise (Pregnancy, puerperium and perinatal conditions) | 1 | 0 — Unrelated
Congenital anomaly (Congenital, familial and genetic disorders) | 1 | 0 — Unrelated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT04547023/Prot_001.pdf
  • Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT04547023/SAP_002.pdf
  • Informed Consent Form (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT04547023/ICF_003.pdf